CLINICAL TRIAL: NCT04678947
Title: The BARF Project: A Pilot Study Using the BARF Scale to Assess CINV in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Original investigator left the university
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202012147
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BARF scale (Experimental): * Nursing staff (which may include patient technicians and nursing assistants) will use the scale to assess the patient's nausea for the entire duration of the admission. These assessments will take place in conjunction with vital sign monitoring, every 4 hours. The associated script will be read while the laminated scale is shown to the patient.
  * The nurse will then log the patient's response in the patient's electronic medical record
  Interventions: Behavioral: Baxter Retching Faces (BARF) scale
- No intervention (No Intervention): -Patients in the control group will proceed with their inpatient chemotherapy admissions without any interventions. These admissions will take place prior to the admissions of the experimental group, so as not to bias providers.

INTERVENTIONS:
Behavioral: Baxter Retching Faces (BARF) scale — * Pictorial scale that was developed for use by pediatric patients in self-reported assessments of nausea severity
  * A patient will respond by choosing a picture or a number on the scale that best represents how they feel. The patient may speak or simply point to their response. While the numbers 0-2-4-6-8-10 are listed alongside the pictures, patients are also allowed to choose "in between" or odd numbers. If a patient is unwilling to participate, the patient's parent or guardian may serve as their proxy and choose a number for them, based off of their symptoms.
  * The BARF scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).
  Arms: BARF scale

SUMMARY:
In this pilot study, the Baxter Retching Faces (BARF) Scale will be used to assess chemotherapy induced nausea and vomiting (CINV) in the pediatric cancer population during chemotherapy admissions, and the corresponding administration of anti-emetic medications will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer of any kind.
* Patients receiving inpatient chemotherapy at SLCH on the general pediatric oncology service
* Patients admitted for a course of inpatient chemotherapy scheduled to last at least 24 hours and but no more than 7 days.
* Patients who have received any prior cancer treatment, including radiation therapy, and/or surgery.
* Patients ages 4 to 12 years of age.
* Patient with a guardian who has the ability to understand English and the willingness to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Any patient who is not undergoing inpatient chemotherapy on the general pediatric oncology service, including patients undergoing chemotherapy as conditioning for hematopoietic stem cell transplantation or other cellular therapy.
* Any patient who is receiving their first cycle of inpatient chemotherapy (however, they can be included during a future cycle).
* Any patient who is blind or unable to communicate by speaking or pointing.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Doses of anti-emetic medication administered during inpatient chemotherapy admissions | 24 hours - 7 days (estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Armstrong, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu